CLINICAL TRIAL: NCT06776653
Title: Impact of a Snoezelen Element on Anxiety in Patients With Special Needs During Oral Care at the Hôtel-Dieu University Hospital in Nantes: A Real-Life Study at Nantes University Hospital
Brief Title: Impact of a Snoezelen Element on Anxiety in Patients During Oral Care: A Real-Life Study at Nantes University Hospital
Acronym: IISLA
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AP_IH_IISLA_01
Record Dates: First submitted 2024-12-20; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Odontologic Disorders
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tovertafel Pixie: Patients who will have the Tovertafel Pixie in the waiting room and the consultation room
  Interventions: Other: Tovertafel Pixie
- controle: Patients without the Tovertafel Pixie in the waiting room and the consultation room

INTERVENTIONS:
Other: Tovertafel Pixie — The Tovertafel Pixie® projector has a distracting effect, which can help divert the patient's attention while waiting for or undergoing treatment.
  Groups: Tovertafel Pixie

SUMMARY:
Research on dental phobia highlights both external causes, like traumatic experiences or media influence, and internal factors, such as genetics and personality traits. While many studies focus on technical aspects of dental care, few explore how the care environment affects patient anxiety.

The Snoezelen concept, developed in the 1970s, uses sensory stimulation (sight, sound, smell, and touch) to reduce anxiety. Initially designed for individuals with neurocognitive disorders, it creates a calming environment and has since been adopted in various healthcare settings.

At Nantes University Hospital, the dental department will test the Tovertafel Pixie®, a sensory projector designed to distract patients and reduce anxiety. Its mobility allows it to be used in waiting rooms and treatment areas, projecting onto ceilings, walls, or tables. This real-life study will assess whether patients exposed to the projector experience less anxiety compared to those who are not, with the goal of improving patient care and dental treatment experiences.

DETAILED DESCRIPTION:
The study involves a questionnaire that the dental department usually provide to our patients, which is partially completed by the patient and partially by the practitioner at the end of the treatment session. No follow-up visit is required.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, over 18 years old;
* consulting in the specialized care unit;
* who understands French;
* receiving care in the specialized dentistry unit and capable of expressing themselves independently regarding the various items in the questionnaire, whether orally, in writing, through a speech synthesis system, or using pictograms;
* able to provide consent to participate.

Exclusion Criteria:

* receiving care in the specialized care unit who are unable to express themselves independently regarding the various items in the questionnaire, whether orally, in writing, through a speech synthesis system, or using pictograms;
* refuse to participate in the study;
* under guardianship, curatorship, or legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients consulting the specialized care unit of the dentistry department at Hôtel-Dieu University Hospital in Nantes, capable of understanding the various questions independently or with the assistance of a trusted person
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Measurement of anxiety. | 1 day
  The Kleinknecht Dental Fear Survey (DFS) measures dental anxiety on a scale ranging from 20 (minimum) to 100 (maximum), where higher scores indicate greater levels of fear or anxiety - Comparison of means

SECONDARY OUTCOMES:
Measure the waiting time in the waiting room | 1day
  Measure the waiting time in the waiting room in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Hyon, M.D, Principal Investigator — Nantes University Hospital

IPD SHARING:
Plan to Share IPD: Undecided